CLINICAL TRIAL: NCT00724334
Title: An Open-Label Study to Evaluate the Long-Term Effects of Orally Administered SAR302503 in Patients With Primary or Secondary Myelofibrosis
Brief Title: A Long-Term Study of the Effects of Orally Administered SAR302503 in Patients With Myelofibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED12015; MF-TG101348-002 (Other: Targegen)
Record Dates: First submitted 2008-07-17; First posted 2008-07-29 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2016-02

CONDITIONS: Myelofibrosis
Keywords: myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SAR302503 (TG101348)

INTERVENTIONS:
Drug: SAR302503 (TG101348) — orally administered, once a day

SUMMARY:
The purpose of this study is to evaluate the long-term effects of orally administered SAR302503 (TG101348) in patients with myelofibrosis who have completed the MF-TG101348-001 study.

DETAILED DESCRIPTION:
SAR302503 (TG101348) is a potent small molecule inhibitor of Janus kinase 2 (JAK2). This is an extension study for a first-in-man, dose escalation study (MF-TG101348-001). The safety, tolerability and clinical activity of SAR302503 (TG101348) in subjects with myelofibrosis will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Completion of MF-TG101348-001 study
* Diagnosis of myelofibrosis
* At least 18 years of age

Exclusion Criteria:

* Any acute or chronic medical abnormality that may increase the risk associated with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety (i.e. adverse events, effects on laboratory parameters, vital signs and ECGs) and tolerability | 6 months

SECONDARY OUTCOMES:
Clinical activity and pharmacodynamics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ayalew Tefferi, MD, Study Chair — Mayo Clinic, Rochester, MN
Locations (6):
- United States (6):
  - Investigational Site Number 840103, La Jolla, California
  - Investigational Site Number 840102, Stanford, California
  - Investigational Site Number 840105, Boston, Massachusetts
  - Investigational Site Number 840106, Ann Arbor, Michigan
  - Investigational Site Number 840104, Rochester, Minnesota
  - Investigational Site Number 840101, Houston, Texas

REFERENCES:
- See also: MPD Foundation — http://mpdfoundation.org/